CLINICAL TRIAL: NCT05296434
Title: Delta Radiomics Based on Gd-EOB-DTPA-enhanced MRI for Quantitative Evaluation of Liver Function
Brief Title: Delta Radiomics for Liver Function Evaluation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Yingfang Fan, Professor, Zhujiang Hospital
Other Study IDs: 2021-KY-105-02
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Chronic Liver Disease
Keywords: liver function; magnetic resonance imaging; radiomics; chronic liver disease; quantitative assement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control Group: Healthy volunteers undergoing MRI exam, ICG test and blood biochemical tests
- Child-Pugh A Group: Composed of patients with liver function of Child-Pugh A grade undergoing MRI exam, ICG test and blood biochemical tests
- Child-Pugh B Group: Composed of patients with liver function of Child-Pugh B grade undergoing MRI exam,ICG test and blood biochemical tests
- Child-Pugh C Group: Composed of patients with liver function of Child-Pugh C grade undergoing MRI exam

SUMMARY:
To evaluate the feasibility and efficacy of delta radiomics-derived index based on Gd-EOB-DTPA enhanced MRI as a new imaging biomarker for the quantitative assessment of liver function.

DETAILED DESCRIPTION:
Delta radiomics is a novel concept proposed on the basis of radiomics. It can be used to evaluate the dynamic changes of imaging features in the time dimension, reflecting functional information of the tissue.

In clinical practice, liver function can be evaluated by gadoxate enhanced MRI by measuring signal intensity. Most often, simple visual assessment is performed, but quantitative measurements are also done. Theoretically, liver function should also be possible to quantify by using delta radiomics, ie by subtracting MR imaging features obtained in the earlier phase from the latter phase.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old, no gender limit.
* Patients with chronic liver disease and different degrees of liver damage (Child-Pugh A, B and C) and healthy controls.
* No history of liver-related surgery (except for cholecystectomy).
* No cardiopulmonary diseases or other diseases which may impair liver function.
* Agree to participate in the study and provide written informed consent.

Exclusion Criteria:

* Alcoholic hepatitis, non-alcoholic fatty liver disease, or autoimmune hepatitis.
* Liver tumors or metastasis or other extraheptic tumor.
* Splenectomy or other cases where the spleen is absent.
* Chronic kidney disease, renal damage.
* Allergy to contrast agents or other conditions that cannot undergo Gd-EOB-DTPA enhanced MRI exam.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and patients with different degrees of liver function impairment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between delta radiomics parameter and ICG test in assessment of liver function | within 3 days
  MRI and ICG tests performed within 3 days apart

SECONDARY OUTCOMES:
Correlation between delta radiomics parameter and serum biochemical tests in assessment of liver function | with 3 days
  MRI and blood biochemical tests performed within 3 days apart

CONTACTS AND LOCATIONS:
Locations (1):
- The First Department of Hepatobiliary Surgery, Zhujiang Hospital, Guangzhou, Guangdong, China